CLINICAL TRIAL: NCT03700970
Title: Double-Blinded Randomized Control Trial Comparing Liposomal Bupivacaine and Bupivacaine Hydrochloride in Transversus Abdominis Plane Blocks Prior To DIEP Flap for Breast Reconstruction
Brief Title: Comparing Local Anesthetics for TAP Block During Abdominally-based Free Flap for Breast Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Galen Perdikis, Chair and Professor of Surgery Department of Plastic Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 180421
Record Dates: First submitted 2018-10-02; First posted 2018-10-09 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Breast Reconstruction; Anesthesia; Transverse Abdominis Plane Block
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and plastic surgeons will be blinded to the study treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAP block with liposomal bupivacaine (Experimental): Local analgesia (TAP blocks) will be administered under ultrasound guidance in the operating room after the patient is intubated and under general anesthesia. Under sterile conditions and ultrasound guidance, the fascial plane between the internal oblique and transversus abdominis muscles (muscles of the abdominal wall) will be identified at the anterior axillary line, midway between the costal margin and iliac crest. The epidural needle will be inserted through the skin to the appropriate fascial plane, and the local anesthetic will be injected in that plane. 20mL of Exparel® 1.3% mixed with 20mL of 0.25% bupivacaine, for a total of 40mL of local anesthestic mixture, 20mL to be injected on each side.
  Interventions: Drug: Liposomal bupivacaine
- TAP block with regular bupivacaine (Active Comparator): Local analgesia (TAP blocks) will be administered under ultrasound guidance in the operating room after the patient is intubated and under general anesthesia. Under sterile conditions and ultrasound guidance, the fascial plane between the internal oblique and transversus abdominis muscles (muscles of the abdominal wall) will be identified at the anterior axillary line, midway between the costal margin and iliac crest. The epidural needle will be inserted through the skin to the appropriate fascial plane, and the local anesthetic will be injected in that plane. 20mL of 0.25% bupivacaine injected on each side.
  Interventions: Drug: Regular bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — 20mL of Exparel® 1.3% mixed with 20mL of 0.25% bupivacaine, for a total of 40mL of local anesthestic mixture, 20mL to be injected on each side.
  Other Names: LB
  Arms: TAP block with liposomal bupivacaine
Drug: Regular bupivacaine — 20mL of 0.25% bupivacaine injected on each side.
  Other Names: Bupivacaine HCl
  Arms: TAP block with regular bupivacaine

SUMMARY:
This study will compare the efficiency of transversus abominus plane (TAP) block using liposomal bupivacaine versus plain bupivacaine that is administered in the operating room under ultrasound guidance prior to the in patients undergoing abdominally-based free flap breast reconstruction at Vanderbilt University Medical Center.

DETAILED DESCRIPTION:
Transversus Abdominis Plane (TAP) blocks are commonly used as part of Enhanced Recovery After Surgery (ERAS) pathway. This prospective, double-blinded, randomized control trial compares post-operative pain and narcotic consumption after deep inferior epigastric artery perforator (DIEP) breast reconstruction with liposomal bupivacaine (LB) compared to bupivacaine hydrochloride (BHCl). Subjects undergoing DIEP flaps were randomly assigned LB or BHCl, performed using ultrasound-guided TAP block technique pre-procedurally. Primary outcomes were postoperative narcotic analgesia required in oral morphine equivalents (OME) from postoperative day (POD) 0 to 7. Secondary outcomes included POD 1-7 pain Numeric Rating Scale (NRS), non-narcotic pain medication consumption, time to first narcotic use, return of bowel function, and length of stay (LOS).

ELIGIBILITY:
Inclusion Criteria:

1. age between 18-85 years
2. males or females
3. plastic surgery for abdominally-based free flap breast reconstruction.

Exclusion Criteria:

1. those not candidates for TAP blocks due to allergies to the medications (e.g., bupivacaine)
2. those with anatomic contra-indications to performing a TAP block
3. those unwilling to participate in follow-up assessments
4. vulnerable populations
5. chronic pain or associated diagnosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galen Perdikis, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen L, Glassman GE, Afshari A, Feng X, Shastri UD, Kaoutzanis C, McEvoy MD, Bansal V, Canlas C, Yao J, Higdon K, Perdikis G. Randomized Controlled Trial Comparing Liposomal to Plain Bupivacaine in the Transversus Abdominis Plane for DIEP Flap Breast Reconstruction. Plast Reconstr Surg. 2024 Mar 1;153(3):543-551. doi: 10.1097/PRS.0000000000010710. Epub 2023 May 22. PMID 37220228

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Started | 30 | 30
Completed | 21 | 19
Not Completed | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Transversus Abdominis Plane (TAP) Block With Liposomal Bupivacaine: Local analgesia (TAP blocks) will be administered under ultrasound guidance in the operating room after the patient is intubated and under general anesthesia. Under sterile conditions and ultrasound guidance, the fascial plane between the internal oblique and transversus abdominis muscles (muscles of the abdominal wall) will be identified at the anterior axillary line, midway between the costal margin and iliac crest. The epidural needle will be inserted through the skin to the appropriate fascial plane, and the local anesthetic will be injected in that plane. 20mL of Exparel® 1.3% mixed with 20mL of 0.25% bupivacaine, for a total of 40mL of local anesthestic mixture, 20mL to be injected on each side.
  Liposomal bupivacaine: 20mL of Exparel® 1.3% mixed with 20mL of 0.25% bupivacaine, for a total of 40mL of local anesthestic mixture, 20mL to be injected on each side.
- Transversus Abdominis Plane (TAP) Block With Regular Bupivacaine: Local analgesia (TAP blocks) will be administered under ultrasound guidance in the operating room after the patient is intubated and under general anesthesia. Under sterile conditions and ultrasound guidance, the fascial plane between the internal oblique and transversus abdominis muscles (muscles of the abdominal wall) will be identified at the anterior axillary line, midway between the costal margin and iliac crest. The epidural needle will be inserted through the skin to the appropriate fascial plane, and the local anesthetic will be injected in that plane. 20mL of 0.25% bupivacaine injected on each side.
  Regular bupivacaine: 20mL of 0.25% bupivacaine injected on each side.
- Total: Total of all reporting groups
Arm/Group | Transversus Abdominis Plane (TAP) Block With Liposomal Bupivacaine | Transversus Abdominis Plane (TAP) Block With Regular Bupivacaine | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (9.5) | 52.2 (9.8) | 52.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (5.3) | 30.2 (4.3) | 29.9 (4.8)
Smoker [Count of Participants; unit: Participants] | 1 | 0 | 1
Diabetic [Count of Participants; unit: Participants] | 8 | 6 | 14
Hypertension (HTN) [Count of Participants; unit: Participants] | 9 | 10 | 19
Hypercoagulable states [Count of Participants; unit: Participants] | 1 | 0 | 1
History of hormonal therapy (HT) [Count of Participants; unit: Participants]
  None | 12 | 17 | 29
  Prior HT | 5 | 3 | 8
  Current HT | 13 | 10 | 23
Prior radiation [Count of Participants; unit: Participants] | 6 | 10 | 16
Immunosuppressive medications [Count of Participants; unit: Participants] | 1 | 1 | 2
Prior chemotherapy [Count of Participants; unit: Participants] | 10 | 10 | 20
Deep Inferior Epigastric Artery Perforator (DIEP) Laterality [Count of Participants; unit: Participants]
  Unilateral DIEP | 9 | 7 | 16
  Bilateral DIEP | 21 | 23 | 44
DIEP timing [Count of Participants; unit: Participants] — DIEP timing is divided as immediate or delayed: "immediate DIEP" refers to reconstruction performed at the same time as the mastectomy and "delayed DIEP" refers to reconstruction performed weeks, months, or years later.
  Participants
    Immediate DIEP | 5 | 6 | 11
    Delayed DIEP | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Amount of Supplemental Postoperative Narcotic Analgesia in Oral Morphine Equivalents (OME)
Description: Amount of supplemental postoperative narcotic analgesia (both intravenous and oral) required by study groups in oral morphine equivalents
Time Frame: Postoperative day (POD) 1 to 7
Measure: Mean (Standard Deviation); unit: mg morphine equivalents
Arm/Group | Transversus Abdominis Plane (TAP) Block With Liposomal Bupivacaine | Transversus Abdominis Plane (TAP) Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
mg morphine equivalents
  POD 1 | 19.8 (18.8) | 23.6 (17.5)
  POD 2 | 20.7 (20.5) | 25.2 (23.5)
  POD 3 | 12.2 (15.3) | 12.8 (11.7)
  POD 4 | 8.2 (8.7) | 8.8 (9.3)
  POD 5 | 7.33 (8.48) | 6.52 (8.51)
  POD 6 | 5.1 (7.0) | 6.8 (7.7)
  POD 7 | 3.8 (5.9) | 4.9 (7.7)

2. Secondary Outcome: Pain Measure
Description: Pain as measured by numeric rating scale ranging from 0 (no pain) to 10 (worst pain ever).
Time Frame: Post operative day (POD) 1 to 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
score on a scale
  POD 1 | 2.43 (1.98) | 2.93 (2.80)
  POD 2 | 2 (1.7) | 3.1 (3)
  POD 3 | 2.9 (2.3) | 3.1 (2.5)
  POD 4 | 2.9 (2.2) | 3.1 (2.7)
  POD 5 | 2.6 (2.2) | 3.1 (2.6)
  POD 6 | 2.3 (2.1) | 3.2 (2.7)
  POD 7 | 2.3 (2.3) | 2.8 (2.5)

3. Secondary Outcome: Time to First Opiate Use
Description: Time from end of surgery to time of first opioid intake measured in hours
Time Frame: 0-29.8 hours post operation
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
hours | 12.4 (17.4) | 8.2 (19.8)

4. Secondary Outcome: Time to Return of Bowel Function
Description: Mean time in days at which patients had a return of bowel movement post op
Time Frame: 1 to 4 days post operation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
days | 2.62 (0.97) | 2.58 (0.97)

5. Secondary Outcome: Length of Stay
Description: Length of hospital stay post operatively
Time Frame: 1 to 4 days
Measure: Mean (Standard Deviation); unit: DAYS
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
DAYS | 2.43 (0.77) | 2.23 (0.43)

6. Secondary Outcome: Ambulation
Description: Time to first ambulate post op (in days)
Time Frame: 1 day post op
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
days | 1 (0) | 1 (0)

7. Secondary Outcome: Non-narcotic Pain Medication Intake: Acetaminophen
Description: The total use of the non-narcotic pain medication Acetaminophen was recorded during hospitalization
Time Frame: Post op day 1 to 7
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
milligrams
  POD 1 | 2630 (803) | 2840 (503)
  POD 2 | 2937 (972) | 2868 (799)
  POD 3 | 2160 (1334) | 1945 (1342)
  POD 4 | 1937 (1239) | 1722 (116)
  POD 5 | 1757 (1159) | 1755 (1130)
  POD 6 | 1903 (1179) | 1755 (1067)
  POD 7 | 1887 (1174) | 1588 (1171)

8. Secondary Outcome: Non Narcotic Pain Medication Intake: Cyclobenzaprine
Description: The total use of the non-narcotic pain medication Cyclobenzaprine was recorded during hospitalization
Time Frame: Post op day 1 to 7
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
milligrams
  POD 1 | 0.5 (1.5) | 1.2 (5.5)
  POD 2 | 2 (4.3) | 1.2 (4.1)
  POD 3 | 2.5 (4.9) | 1.5 (4.4)
  POD 4 | 3.7 (8.1) | 1.7 (4.8)
  POD 5 | 3.7 (7.2) | 1.8 (4.8)
  POD 6 | 4 (8.3) | 1.8 (4.8)
  POD 7 | 3 (6.8) | 2.2 (5)

9. Secondary Outcome: Non Narcotic Pain Medication Intake: Gabapentin
Description: The total use of the non-narcotic pain medication gabapentin was recorded during hospitalization
Time Frame: Post op day 1 to 7
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
milligrams
  POD 1 | 730 (315) | 750 (298)
  POD 2 | 807 (358) | 813 (356)
  POD 3 | 680 (489) | 577 (378)
  POD 4 | 603 (454) | 517 (371)
  POD 5 | 537 (451) | 583 (397)
  POD 6 | 503 (453) | 560 (443)
  POD 7 | 457 (449) | 527 (445)

10. Secondary Outcome: Non Narcotic Pain Medication Intake: Celebrex
Description: The total use of the non-narcotic pain medication celebrex was recorded during hospitalization
Time Frame: post op day 1 to 7
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
milligrams
  POD 1 | 200 (144) | 187 (138)
  POD 2 | 193 (146) | 203 (119)
  POD 3 | 67 (132) | 60 (113)
  POD 4 | 20 (61) | 0 (0)
  POD 5 | 20 (61) | 0 (0)
  POD 6 | 13 (51) | 0 (0)
  POD 7 | 13 (51) | 0 (0)

11. Secondary Outcome: Non Narcotic Pain Medication Intake: Ondansetron
Description: The total use of the non-narcotic pain medication ondansetron was recorded during hospitalization
Time Frame: Post op day 1 to 7
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
Number analyzed (Participants) | 30 | 30
milligrams
  POD 1 | 1.3 (2.6) | 2.3 (3.3)
  POD 2 | 0.4 (1.6) | 0.4 (1.2)
  POD 3 | 0.27 (1.46) | 0.27 (1.01)
  POD 4 | 0 (0) | 0 (0)
  POD 5 | 0 (0) | 0 (0)
  POD 6 | 0 (0) | 0 (0)
  POD 7 | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TAP Block With Liposomal Bupivacaine | TAP Block With Regular Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAP Block With Liposomal Bupivacaine (N=30) | TAP Block With Regular Bupivacaine (N=30)
Bupivacaine toxicity (Blood and lymphatic system disorders) | 0 | 0
Narcotic complication (Blood and lymphatic system disorders) | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0
Flap loss (Skin and subcutaneous tissue disorders) | 0 | 0

LIMITATIONS AND CAVEATS:
If a patient was unable to be reached, they were given a log to record pain scores and medication intake. There may be a recall bias if those patients were unable to adhere to the protocol to record daily and retroactively logged their scores and number of tablets taken. Another limitation is the reliance of certain outcomes on subjective data (i.e. Numeric Pain Scale scores).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03700970/Prot_001.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03700970/SAP_002.pdf
  • Informed Consent Form (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03700970/ICF_000.pdf